CLINICAL TRIAL: NCT03998007
Title: Development of a Medical Device Utilizing an EEG-Based Algorithm for the Objective Quantification of Pain
Status: Completed | Type: Observational
Sponsor: PainQx, Inc (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 00001
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: IRIS System — A QEEG based pain biomarker that scales with the patient reported NRS

SUMMARY:
Obtained 19 lead EEG data from 50 chronic pain patients along with their clinical history and self-reported pain scored. Machine learning was used to analyze the EEG data and derive a chronic pain biomarker.

ELIGIBILITY:
Inclusion Criteria:

* Male and female chronic pain patients
* Patients between the ages of 18-85 years
* Patients exhibiting the presence of symptoms in excess of 3 months duration
* Patients suffering from neuropathic (e.g., lower back pain), osteoarthritis, or muscular skeletal pain
* Patients with evidence of pathology related to the painful condition on which diagnosis was made (e.g., results of imaging or diagnostic pain code)
* Patients with NRS pain scores across the full range (1-10) at the time of testing

Exclusion Criteria:

* Patients with medically diagnosed psychotic illness
* Patients with medically diagnosed drug or alcohol dependence in the past 12 months
* Patients with a medical history of head injury with loss of consciousness and amnesia (within the last 2 years)
* Patients with skull abnormalities that preclude the proper placement of the electrodes for the EEG data acquisition
* Patients who have a spinal cord stimulator, or other implantable devices
* Patients for whom the source of pain at the time of the evaluation is associated with: neurological disorders (multiple sclerosis, Parkinson, dementia), diabetes, migraines, or those with reflex / sympathetic dystrophy disorder/complex regional pain syndrome, fibromyalgia, or visceral pain
* Patients with cancer
* Patients on workers compensation or disability
* Patient on anticonvulsant medication
* Patients who have a history of seizures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty (50) male and female pain patients with symptoms in excess of 3 months duration (per the IASP definition of Chronic Pain) between the ages of 18-85 years were enrolled. Subjects who met the inclusion/exclusion criteria were asked to volunteer for the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Pearsons Correlation between IRIS derived pain biomarker and patient reported Numeric Rating Scale (0-10) | 6 Months
  A Pearson Correlation of 1.0 is perfection correlation and 0 no correlation between the two measured variables

CONTACTS AND LOCATIONS:
Overall Officials: William Koppes, Principal Investigator — PainQx, Inc
Locations (1):
- Boston Pain Care Center, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided